CLINICAL TRIAL: NCT02853253
Title: Rate of Bronchopulmonary Dysplasia in Preterms Neonates Less Than 29 Weeks' Gestational Age and / or With Birth Weight Less Than 1000 g: a Double Blind Randomized Controlled Multicenter Trial Comparing SMOFlipid and Medialipide
Brief Title: Rate of Bronchopulmonary Dysplasia in Preterms Neonates: a Trial Comparing SMOFlipid and Medialipide
Acronym: SMOF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: scientific question reconsidered
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL16_0135
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Preterm Neonates
Keywords: Preterm neonates
MeSH Terms: interventions — SMOFlipid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMOF (Experimental): parenteral nutrition using SMOFlipid® (FreseniusKabi France, Sèvres, France)
  Interventions: Dietary Supplement: SMOFlipid®
- Medialipide® (Active Comparator): parenteral nutrition using Medialipide® 20% (B Braun Medical, Boulogne, France)
  Interventions: Dietary Supplement: Medialipide®

INTERVENTIONS:
Dietary Supplement: SMOFlipid® — SMOFlipid® (FreseniusKabi France, Sèvres, France). It is a 3rd generation LE containing a physical mixture of soybean oil (30%), MCT (30%), olive oil (25%) and fish oil (15%). Its ratio omega6/omega 3 is 2,5/1. SMOF will be initiated within the 1st day of life of neonates and will be prescribed daily by the attending physician following these guidelines: initiation rate: 1 g/kg/day; daily increase: 0.5 to 1 g/kg/day ; target: 3 to 4 g/kg/day.
  All included preterms will receive nutritional support according to a single protocol based on the ESPGHAN recommendations: parenteral glucose and amino acids (Primene 10%, Clintec Parenteral, Maurepas, France) soon after birth (in their 1st day of life). Initiation rate of parenteral glucose and amino acids will be 6 to 8 g/kg/day and 2 g/kg/day respectively. The daily increase of parenteral glucose and amino acids will be 1 to 2 g/kg/day and 0.5 g/kg/day respectively, for a target rate of 14 to 17 g/kg/day and 3.5 g/kg/day respectively.
  Arms: SMOF
Dietary Supplement: Medialipide® — Medialipide® 20% (B Braun Medical, Boulogne, France). It is a second generation LE containing soybean oil (50%) and MCT (50%). Its ratio omega6/omega 3 is 7/4. Medialipide will be initiated within the 1st day of life of neonates and will be prescribed daily by the attending physician following these guidelines: initiation rate: 1 g/kg/day ; daily increase: 0.5 to 1 g/kg/day; target: 3 to 4 g/kg/day.
  All included preterms will receive nutritional support according to a single protocol based on the ESPGHAN recommendations: parenteral glucose and amino acids (Primene 10%, Clintec Parenteral, Maurepas, France) soon after birth (in their 1st day of life). Initiation rate of parenteral glucose and amino acids will be 6 to 8 g/kg/day and 2 g/kg/day respectively. The daily increase of parenteral glucose and amino acids will be 1 to 2 g/kg/day and 0.5 g/kg/day respectively, for a target rate of 14 to 17 g/kg/day and 3.5 g/kg/day respectively.
  Arms: Medialipide®

SUMMARY:
SMOF is a large double blind placebo-controlled randomized clinical trial aiming to compare the rate of bronchopulmonary dysplasia (BPD) at 36 weeks corrected age in premature infants < 29 weeks and / or with birth weight < 1000 g receiving either SMOFlipid® or Medialipide® 20%. This study will offer new information for optimizing the management of preterms requiring parenteral nutrition. The investigators hypothesis is that the composition of SMOFlipid may decrease lipid peroxidation and oxidative stress in preterms, resulting in a lower incidence of BPD.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with gestational age < 29 weeks and / or birth weight < 1000 g
* Admission in the Intensive Care Unit within 6 h after birth
* IV Lipid Emulsion (LE) started latest at first day of life
* Anticipated duration of Parenteral Nutrition >10 days
* Informed consent from legal representative

Exclusion Criteria:

* Inherited metabolic diseases
* Major congenital malformations
* Participation to another study evaluating any kind of medications

Ages: 6 Hours to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Rate of other free radical diseases | 36 weeks corrected age
  Free radical diseases include: intraventricular hemorrhage (IVH) > grade II, retinopathy of prematurity (ROP) > grade II, and necrotizing enterocolitis (NEC) > grade IA (Bell classification).

SECONDARY OUTCOMES:
Weight gain | at day 28
  Weight gain in g/kg/j according to the following formulae: 1000 * ((weight on day 28 or week 36 - birth weight)/((weight on day 28 or week 36 + birth weight)/2)) / number of days
Weight gain | week 36 corrected age
  Weight gain in g/kg/j according to the following formulae: 1000 * ((weight on day 28 or week 36 - birth weight)/((weight on day 28 or week 36 + birth weight)/2)) / number of days
Growth velocity | at day 28
  Length growth velocity in cm/week at day 28 according to the following formulae: (length on day 28 - length at birth) / number of weeks
Growth velocity | week 36 corrected age
  Length growth velocity in cm/week at week 36 corrected age according to the following formulae: (length on week 36 - length at birth) / number of weeks
Head circumference growth velocity | at day 28
  Head circumference growth velocity in cm/week according to the following formulae: (head circumference on day 28 - head circumference at birth) / number of weeks
Head circumference growth velocity | at week 36 corrected age
  Head circumference growth velocity in cm/week according to the following formulae: (head circumference on week 36 - head circumference at birth) / number of weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CLARIS, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No